CLINICAL TRIAL: NCT05437913
Title: Brief Self-Compassion Intervention for Adolescents With Diabetes Type 1 and Their Caregivers: Protocol for a Single Case Multiple-baseline Feasibility Study
Brief Title: Protocol for Self-Compassion Intervention for Teens With Diabetes Type 1 and Their Caregivers
Acronym: SWEET
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Valencia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: SWEET2021
Record Dates: First submitted 2021-10-13; First posted 2022-06-29 (Actual); Last update posted 2022-06-29 (Actual); Status verified 2021-11

CONDITIONS: Diabetes type1
MeSH Terms: interventions — Psychosocial Intervention

STUDY DESIGN:
Intervention Model Description: single case multiple randomized baseline design
Masking Description: No blinding can be used however the researcher will be blinded when coding observational data.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Self compassion intervention (Other): 4 weeks group and online format self compassion intervention
  Interventions: Other: Psychological intervention (self-compassion based)

INTERVENTIONS:
Other: Psychological intervention (self-compassion based) — 4 weeks intervention for both primary caregivers and adolescents with T1D will be done online through videoconferencing and will be based on three validated protocols that use self-compassion (MSC and MSC Teens).

SUMMARY:
The goal of this study is to examine the feasibility and potential effectiveness of a short (4 sessions) self-compassion intervention for adolescents with T1D and their caregivers on psychological, metabolic, and behavioral outcomes.

DETAILED DESCRIPTION:
Type 1 Diabetes (TD1) has a significant impact on individuals dealing with this chronic metabolic condition, their families and the whole society. A particularly vulnerable group of individuals with TD1 are adolescents. The investigators created a short (4 sessions) self-compassion intervention for adolescents with T1D and their caregivers. Both feasibility and potential clinical effectiveness will be assessed using a single-case, multiple baseline experimental design where psychological, behavioral, and metabolic outcomes will be evaluated at baseline, post intervention, and 3- and 6-months follow ups. Moreover, ecological momentary assessment will be performed daily.

ELIGIBILITY:
Inclusion Criteria for the caregivers:

* have taken care of the management of the patient with diabetes for at least one year since the day of recruitment
* they have access to a personal mobile phone.

Inclusion Criteria for the patients/teens:

* aged 11-15 years old
* diagnosed with T1D more than 12 months ago at the time of recruitment
* they have access to a personal mobile phone.

General Exclusion Criteria:

* non-Spanish native speakers
* presenting developmental or attention deficit disorders (e.g., autism spectrum disorder, ADHD)
* being diagnosed with a serious mental disorder requiring ongoing treatment (e.g., psychosis) or receiving a pharmacological intervention (e.g., depression, anxiety).

Exclusion criteria for teens:

* untreated hypothyroidism
* recently (in previous 48 hours of the recruiting process) diagnosed with (a) diabetic ketoacidosis (DKA) or (b) severe hypoglycaemia.

Ages: 12 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 8 (Actual)
Dates: Start 2021-09-06 (Actual); Primary Completion 2022-03-15 (Actual); Study Completion 2022-09-15 (Estimated)

PRIMARY OUTCOMES:
Change in Self-report psychological variables: depression (caregivers ) | change in PHQ from pre (Day 1) to post (Day 30). Change in PHQ from post (Day30) to Follow up3 (Month 3). Change in PHQ from Follow up 3 (month 3) to Follow up6 (Month 6)
  - 2 items for caregivers: PHQ-2 (Kroenke, 2003; Spanish version: Wulsin et al., 2002)
Change in Self-report psychological variables: depression ( teens) | change in PHQ from pre (Day 1) to post (Day 30). Change in PHQ from post (Day30) to Follow up3 (Month 3). Change in PHQ from Follow up 3 (month 3) to Follow up6 (Month 6)
  - 2 items for teens: PHQ-2 (Richardson et al., 2010; Spanish version: Arrieta et al., 2017)
Change in Self-report psychological variables: self-compassion (caregivers) | Change in SOCS-S from pre (Day 1) to post (Day 30). Change in SOCS-S from post (Day 30) to follow up3 (Month 3). Change in SOCS-S from follow up 3 (month 3) to follow up 6 (month 6).
  - 20 items for caregivers: SOCS-S (Gu et al., 2020); Spanish version back forward translation
Change in Self-report psychological variables: self-compassion (teens) | Change in SOCS-S from pre (Day 1) to post (Day 30). Change in SOCS-S from post (Day 30) to follow up3 (Month 3). Change in SOCS-S from follow up 3 (month 3) to follow up 6 (month 6).
  - 20 items for teens: SOCS-S (Gu et al., 2020); Spanish version back forward translation and adapted to teens
change in Self-report psychological variables: self-criticism (caregivers) | Change in FSCRS-SR from pre (Day 1) to post (Day 30). Change in FSCRS-SR from post (Day 30) to follow up3 (Month 3). Change in FSCRS-SR from follow up 3 (month 3) to follow up 6 (month 6).
  - 14 items for caregivers: FSCRS-SR (Gilbert, Clarke, Hempel, Miles & Irons, 2004); Spanish version back forward translation
Change in Self-report psychological variables: self-criticism (teens) | Change in FSCRS-SR from pre (Day 1) to post (Day 30). Change in FSCRS-SR from post (Day 30) to follow up3 (Month 3). Change in FSCRS-SR from follow up 3 (month 3) to follow up 6 (month 6).
  - 14 items for teens: FSCRS-SR (Gilbert, Clarke, Hempel, Miles & Irons, 2004); Spanish version back forward translation and adapted to teens
Change in Self-report psychological variables: self care (caregivers) | Change in B-MSC from pre (Day 1) to post (Day 30). Change in B-MSC from post (Day 30) to follow up3 (Month 3). Change in B-MSC from follow up 3 (month 3) to follow up 6 (month 6).
  - 24 items for caregivers: B-MSC (Cook-Cottone, 2018); Spanish version back forward translation
Change in Self-report psychological variables: self care (teens) | Change in B-MSC from pre (Day 1) to post (Day 30). Change in B-MSC from post (Day 30) to follow up3 (Month 3). Change in B-MSC from follow up 3 (month 3) to follow up 6 (month 6).
  - 24 items for teens: B-MSC (Cook-Cottone, 2018); Spanish version back forward translation and adapted to teens
Change in Self-report psychological variables: interoceptive awareness (caregivers) | Change in MAIA-2 from pre (Day 1) to post (Day 30). Change in MAIA-2 from post (Day 30) to follow up3 (Month 3). Change in MAIA-2 from follow up 3 (month 3) to follow up 6 (month 6).
  - 32 items for caregivers: MAIA-2 (Mehling et al., 2018); Spanish version back forward translation
Change in Self-report psychological variables: interoceptive awareness (teens) | Change in MAIA-2 from pre (Day 1) to post (Day 30). Change in MAIA-2 from post (Day 30) to follow up3 (Month 3). Change in MAIA-2 from follow up 3 (month 3) to follow up 6 (month 6).
  - 32 items for teens: MAIA-Y (Joenes et al., 2020); Spanish version back forward translation and adapted to teens

SECONDARY OUTCOMES:
change in metabolic outcome 1 (only teens) | Change in HbA1c from pre (Day 1) to post (Day 30). Change in HbA1c from post (Day 30) to follow up3 (Month 3). Change in HbA1c from follow up 3 (month 3) to follow up 6 (month 6).
  glycated hemoglobin (HbA1c)
change in metabolic outcome 2 (only teens) | Change in TiR from pre (Day 1) to post (Day 30). Change in TiR from post (Day 30) to follow up3 (Month 3). Change in TiR from follow up 3 (month 3) to follow up 6 (month 6).
  continuous glucose monitoring (time in range: TiR)
Change in Self-report diabetes-related variables: diabetes-specific emotional distress (caregivers) | Change in PAID-P from pre (Day 1) to post (Day 30). Change in PAID-P from post (Day 30) to follow up3 (Month 3). Change in PAID-P from follow up 3 (month 3) to follow up 6 (month 6).
  - 14 items: PAID-P (Shapiro et al., 2018); Spanish version back forward translation
Change in Self-report diabetes-related variables: diabetes-specific emotional distress (teens) | Change in PAID-T from pre (Day 1) to post (Day 30). Change in PAID-T from post (Day 30) to follow up3 (Month 3). Change in PAID-T from follow up 3 (month 3) to follow up 6 (month 6).
  - 14 items: PAID-T (Shapiro et al., 2018);Spanish version back forward translation and adapted to teens
Change in Self-report diabetes-related variables: the diabetes family conflict scale (caregivers) | Change in DFCS from pre (Day 1) to post (Day 30). Change in DFCS from post (Day 30) to follow up3 (Month 3). Change in DFCS from follow up 3 (month 3) to follow up 6 (month 6).
  - 8 items: DFCS for caregivers, Hood et al., 2007; Spanish version back forward translation
Change in Self-report diabetes-related variables: the diabetes family conflict scale (teens) | Change in DFCS from pre (Day 1) to post (Day 30). Change in DFCS from post (Day 30) to follow up3 (Month 3). Change in DFCS from follow up 3 (month 3) to follow up 6 (month 6).
  - 8 items: DFCS for teens, Hood et al., 2007; Spanish version back forward translation
Change in Self-report diabetes-related variables: parental report on teen's health-related quality of life | Change in KIDSCREEN-10 from pre (Day 1) to post (Day 30). Change in KIDSCREEN-10 from post (Day 30) to follow up3 (Month 3). Change in KIDSCREEN-10 from follow up 3 (month 3) to follow up 6 (month 6).
  - 10 items: KIDSCREEN-10 (Ravens-Sieberer et al., 2005); Spanish version provided by the same authors
Change in observational behavioural variable (caregiver-teen dyad) | Change in PCIM between pre (Day 1) and post (Day 30).
  caregiver-adolescent dyadic interaction analysis of neutral and conflictual topic discussion based on Holmbeck et al. (2013) Parent-child interaction macro coding manual (PCIM)
Change in ecological momentary assessment: affect (caregivers) | Change between baseline (Day 1-Day11) and post (Day 30-Day 34). Change between post (Day 30-Day 34) and follow up3 (Day 90-Day 104). Change between follow up3 (Day 90-Day 104) and follow up6 (Day 180- Day194).
  - 1 item: created by the research team measure of affect sent once per day to participants
Change in ecological momentary assessment: affect (teens) | Change between baseline (Day 1-Day11) and post (Day 30-Day 34). Change between post (Day 30-Day 34) and follow up3 (Day 90-Day 104). Change between follow up3 (Day 90-Day 104) and follow up6 (Day 180- Day194).
  - 1 item: created by the research team measure of affect sent once per day to participants
Change in ecological momentary assessment self kindness (caregivers ) | Change between baseline (Day 1-Day11) and post (Day 30-Day 34). Change between post (Day 30-Day 34) and follow up3 (Day 90-Day 104). Change between follow up3 (Day 90-Day 104) and follow up6 (Day 180- Day194).
  - 1 item: created by the research team measure of self kindness sent once per day to participants
Change in ecological momentary assessment self kindness (teens) | Change between baseline (Day 1-Day11) and post (Day 30-Day 34). Change between post (Day 30-Day 34) and follow up3 (Day 90-Day 104). Change between follow up3 (Day 90-Day 104) and follow up6 (Day 180- Day194).
  - 1 item: created by the research team measure of self kindness sent once per day to participants
Change in ecological momentary assessment: self criticism (caregivers) | baseline (Day 1-Day11), post (Day 30-Day 34), follow up3 (Day 90-Day 104), and follow up6 (Day 180- Day194)
  - 1 item: created by the research team measure of self criticism sent once per day to participants
Change in ecological momentary assessment: self criticism (teens) | Change between baseline (Day 1-Day11) and post (Day 30-Day 34). Change between post (Day 30-Day 34) and follow up3 (Day 90-Day 104). Change between follow up3 (Day 90-Day 104) and follow up6 (Day 180- Day194).
  - 1 item: created by the research team measure of self criticism sent once per day to participants
Change in ecological momentary assessment: triggering event (caregivers) | Change between baseline (Day 1-Day11) and post (Day 30-Day 34). Change between post (Day 30-Day 34) and follow up3 (Day 90-Day 104). Change between follow up3 (Day 90-Day 104) and follow up6 (Day 180- Day194).
  - 1 item: created by the research team measure of triggering events where the participants are asked to rate how much a potential negative triggering event affected them. The item was sent once per day to participants
Change in ecological momentary assessment: triggering event (teens) | Change between baseline (Day 1-Day11) and post (Day 30-Day 34). Change between post (Day 30-Day 34) and follow up3 (Day 90-Day 104). Change between follow up3 (Day 90-Day 104) and follow up6 (Day 180- Day194).
  - 1 item: created by the research team measure of triggering events where the participants are asked to rate how much a potential negative triggering event affected them. The item was sent once per day to participants
Change in ecological momentary assessment: emotion regulation (caregivers ) | Change between baseline (Day 1-Day11) and post (Day 30-Day 34). Change between post (Day 30-Day 34) and follow up3 (Day 90-Day 104). Change between follow up3 (Day 90-Day 104) and follow up6 (Day 180- Day194).
  - 1 item: created by the research team measure of emotion regulation strategies where the participants are asked to chose from the list emotion regulation strategies that they used to regulate the emotions related to the triggering event. The item was sent once per day to participants
Change in ecological momentary assessment: emotion regulation (teens) | Change between baseline (Day 1-Day11) and post (Day 30-Day 34). Change between post (Day 30-Day 34) and follow up3 (Day 90-Day 104). Change between follow up3 (Day 90-Day 104) and follow up6 (Day 180- Day194).
  - 1 item: created by the research team measure of emotion regulation strategies where the participants are asked to chose from the list emotion regulation strategies that they used to regulate the emotions related to the triggering event. The item was sent once per day to participants
change in ecological momentary assessment: positive impact on caregiver-teen interactions (caregivers and teens) | Change between baseline (Day 1-Day11) and post (Day 30-Day 34). Change between post (Day 30-Day 34) and follow up3 (Day 90-Day 104). Change between follow up3 (Day 90-Day 104) and follow up6 (Day 180- Day194).
  - 1 item: created by the research team measure of positive impact on parent child interaction where the participants are asked to rate how the triggering event impacted their relationship with (caregiver or child) positively. The item was sent once per day to participants
change in ecological momentary assessment: negative impact on caregiver-teen interactions (caregivers and teens) | Change between baseline (Day 1-Day11) and post (Day 30-Day 34). Change between post (Day 30-Day 34) and follow up3 (Day 90-Day 104). Change between follow up3 (Day 90-Day 104) and follow up6 (Day 180- Day194).
  - 1 item: created by the research team measure of positive impact on parent child interaction where the participants are asked to rate how the triggering event impacted their relationship with (caregiver or child) negatively. The item was sent once per day to participants
Practice frequency | during the intervention (Day11-Day 30)
  - 1 item: created by the research team measure of frequency of daily meditation practice
Possible adverse effects | Change between post (Day 30-Day 34) and follow up3 (Day 90-Day 104). Change between follow up3 (Day 90-Day 104) and follow up6 (Day 180- Day194).
  6 item scale developped by the team

CONTACTS AND LOCATIONS:
Overall Officials: Rosa Baños Rivera, PhD, Principal Investigator — Univeristy of Valencia
Locations (1):
- University of Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No